CLINICAL TRIAL: NCT04527094
Title: Development and Prospective Evaluation of a Machine Learning Model to Predict Postoperative Respiratory Failure
Brief Title: Machine Learning Model to Predict Postoperative Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Kyu Yoon, clinical assistant professor, Seoul National University Hospital
Other Study IDs: AI_PRF
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Noncardiac Surgery
Keywords: Artificial Intelligence; Risk Factors; Postoperative respiratory failure; Validation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AI_PRF: Adults patients undergoing general anesthesia
  Interventions: Diagnostic Test: Prediction of postoperative respiratory failure using a machine learning

INTERVENTIONS:
Diagnostic Test: Prediction of postoperative respiratory failure using a machine learning — The performance of a machine learning model to predict postoperative respiratory failure after general anesthesia within postoperative day 7 was tested prospectively.

SUMMARY:
The main objective of this study is to develop a machine learning model that predicts postoperative respiratory failure within 7 postoperative day using a real-world, local preoperative and intraoperative electronic health records, not administrative codes.

DETAILED DESCRIPTION:
Postoperative pulmonary complications are known to increase the length of hospital stay and healthcare cost. One of the most serious form of these complications is postoperative respiratory failure, which is also associated with morbidity and mortality. A lot of risk stratification models have been developed for identifying patients at increased risk of postoperative respiratory failure. However, these models were built by using a traditional logistic regression analysis. A logistic regression analysis had disadvantages of assuming the relationship between dependent and independent variables as linear. Recent advances in artificial intelligence make it possible to manage and analyze big data. Prediction model using a machine learning technique and large-scale data can improve the accuracy of prediction performance than those of previous models using traditional statistics. Furthermore, a machine learning technique may be a useful adjuvant tool in making clinical decisions or real-time prediction if it is integrated into the healthcare system. However, to our knowledge, there was no study investigating the predictive factors of postoperative respiratory failure using a machine-learning approach. Therefore, the main objective of this study is to develop a machine learning model that predicts postoperative respiratory failure within 7 postoperative day using a real-world, local preoperative and intraoperative electronic health records, not administrative codes and evaluate its performance prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients undergoing general anesthesia for noncardiac surgery

Exclusion Criteria:

* Age under 18 years
* Surgery duration < 1 hr
* Cardiac surgery
* Surgery performed only regional or local anesthesia, peripheral nerve block, or monitored anesthesia care
* Organ transplantation
* Patient with preoperative tracheal intubation
* Patients who had tracheostoma prior to surgery
* Patients scheduled for tracheostomy
* Surgery performed outside the operating room
* Length of hospital stay < 24 h

If the patients had multiple surgeries during the same hospital stays, we included the first surgical cases in the dataset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing general anesthesia for noncardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 22250 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
the incidence of postoperative respiratory failure after general anesthesia | within postoperative day 7
  Postoperative respiratory failure which was defined as mechanical ventilation >48 h or any reintubation after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hyun-Kyu Yoon, Seoul, South Korea